CLINICAL TRIAL: NCT06969183
Title: A Descriptive Exploration of Flourishing Through Kink
Status: Completed | Type: Observational
Sponsor: The Alternative Sexualities Health Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: T2024-01
Record Dates: First submitted 2025-02-21; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Impact on Psychological Well-being of Involvement in Kink Behaviors
Keywords: kink, BDSM, flourishing, trauma recovery

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study examines the experiences of people who have engaged in alternative sexual behaviors, like kink or BDSM, and whether there have been any positive effects on well-being

DETAILED DESCRIPTION:
The study design is an observational, cross-sectional mixed methods study with data collected anonymously online via a computer-assisted survey through Qualtrics. Subjects will be recruited through nonprobability snowball sampling

ELIGIBILITY:
Inclusion Criteria:

- 1. Age of majority in the legal jurisdiction (geographic location) where the survey is taken (usually age 18) 2. Self-reported involvement in kink behaviors 3. self-reported English-language proficiency sufficient to understand the study instrument.

4. Answer correctly a series of questions to screen for bots and fraudulent responses

Exclusion Criteria:

* 1. Report no involvement in kink activities or behaviors 2. Answer incorrectly three or more questions for bot detection and fraudulent responses, 3+ out of 4 bot detection questions.

  3. Clearly fraudulent use of the internet survey, such as: evidence of non-human data entry via an internet "bot", duplicative or prank data entry that entails contradictory or clearly fraudulent data.

  4. Any condition that, in the professional judgment of the Principal Investigator, should exclude an individual from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have engaged in kink behaviors
Sampling Method: Non-Probability Sample
Enrollment: 1131 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Reports of Healing through Kink | Baseline
  Primary Outcome measure: the proportion of people who affirmatively answer "Have you ever experienced healing from trauma through kink?"

SECONDARY OUTCOMES:
Subgroups More Likely | Baseline
  Secondary Objective 1: demographic characteristics including gender identity, sexual orientation, yearly household income, yearly individual income, age, racial and ethnic identity, age of involvement in kink behavior and first awareness of kink fantasy/desire; aspects of kink identity
Types of Trauma Involved | Baseline
  Secondary Objective 2: scores on the Life Events Checklist-5, comparing people who have experienced healing through kink to people who have not experienced healing through kink
Attachment Differences | Baseline
  Secondary Objective 3: scores on the Adult Attachment Scale, comparing people who have experienced healing through kink to people who have not experienced healing through kink
Healing and Flourishing | Baseline
  Secondary Objective 4: scores on the Diener Flourishing Scale, comparing people who have experienced healing through kink to people who have not experienced healing through kink
Conditions for Healing through Kink | Baseline
  Secondary Objective 5: responses to questions about kink activities; descriptions of negotiation, aftercare, and debriefing in relation to kink scenes; engagement in professional therapy, comparing people who have experienced healing through kink to people who have not experienced healing through kink
AEDP Features of Healing through Kink | Baseline
  Secondary Objective 6: study will create a measure of features of experience that align with Accelerated Experiential Dynamic Psychotherapy, including keyword analysis of write-in answers for healing experiences; coding variables into a fidelity index of the clinical features of AEDP to reduce measurement error in the constituent AEDP feature variables; correlational and predictive analyses between and among AEDP clinical features/strategies, kink activities, and healing/flourishing scale scores
Level of current symptoms of Trauma | Baseline
  Secondary Objective 7: scores on the PTSD Checklist-5, comparing people who have experienced healing through kink to people who have not experienced healing through kink
Flourishing | Baseline
  Secondary Objective 8: scores on the Flourishing Index, comparing people who have experienced healing through kink to people who have not experienced healing through kink

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Sprott, PhD, Principal Investigator — The Alternative Sexualities Health Research Alliance
Locations (1):
- TASHRA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
anonymity in data collection, no individual participant data will be shared

REFERENCES:
- See also: Website of community based research organization — https://www.tashra.org